CLINICAL TRIAL: NCT05265845
Title: Using Digital Health Technologies to Prevent Rapid Infant Weight Gain.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI transferred to a different institution prior to starting the intervention.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: Pro00109854
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Breastfeeding; Bottle Feeding; Child Obesity
MeSH Terms: conditions — Breast Feeding; Bottle Feeding; Pediatric Obesity | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Interactive text messages that include goal setting, tailored feedback, and skills training.
  Interventions: Behavioral: Intervention
- Control (Active Comparator): Text4Baby
  Interventions: Behavioral: Text4Baby

INTERVENTIONS:
Behavioral: Intervention — The intervention aims to support infant feeding decisions and teach responsive feeding strategies.
  Arms: Intervention
Behavioral: Text4Baby — Free health and wellness text messages timed to due date through pregnancy and up until the baby's first birthday.
  Arms: Control

SUMMARY:
A digital intervention to provide supplemental infant feeding support to mothers enrolled in WIC. The trial begins prenatally and continues through 3-months postpartum and tests the feasibility and acceptability of a text messaging intervention aimed at increasing responsive bottle feeding as well as breastfeeding duration and exclusivity among mothers enrolled in WIC using evidence-based components such as interactive self-monitoring and feedback.

Recruitment and enrollment never started at Duke for the Intervention represented in this record. The overall status of recruiting and actual start date were previously entered in error.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in WIC, English or Spanish speaking, at least 18 years old, between 18-28 weeks' gestation, and planning to remain enrolled in WIC for 6 months, intention to breastfeed or undecided about breastfeeding, and willingness to send and receive daily text messages.

Exclusion Criteria:

* Postpartum exclusions include infant prematurity (<37 weeks), >3 days in neonatal intensive care unit, major medical problem affecting breastfeeding (i.e., maternal HIV), or birth weight <5 lbs.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Engagement | 32 weeks gestation to 3 months postpartum
  Percent of text messages responded to as measured by text log.

SECONDARY OUTCOMES:
Breastfeeding duration | 0 to 3 months postpartum
  Number of weeks breastfed as measured by patient response.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa C Kay, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center - with Piedmont Health Services, Inc., Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No